CLINICAL TRIAL: NCT00003843
Title: UGT1A1 Polymorphism in Patients With Colorectal Cancer Treated With CPT-11 (Irinotecan)
Brief Title: Irinotecan in Treating Patients With Colorectal Cancer
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to poor accrual
Sponsor: California Cancer Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000067003; LAC-USC-3C981; NCI-G99-1513
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2013-09

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Irinotecan; Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Drug: irinotecan hydrochloride
Genetic: mutation analysis
Genetic: polymorphism analysis

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irinotecan in treating patients who have colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency of genetic polymorphisms of UGT1 in Hispanics with colorectal cancer.
* Determine if pharmacokinetics of irinotecan and its metabolites, SN38 and SN38G, are associated with the genotype of UGT1 and clinical toxicity.
* Determine whether the genetic polymorphisms of UGT1 are associated with clinical toxicity and pharmacokinetics/pharmacodynamics of irinotecan in patients with unresectable colorectal cancer treated with irinotecan.
* Determine the response, time to progression, and survival in patients with UGT1A1 polymorphisms treated with irinotecan.

OUTLINE: Genomic DNA is isolated from blood samples from patients and analyzed for UGT1 polymorphisms. Patients are stratified according to UGT1 genotype (homozygous for wild type vs heterozygous for abnormal allele vs homozygous for abnormal allele).

Patients receive irinotecan over 90 minutes weekly for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: Approximately 28 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven advanced or disseminated colorectal cancer

  * Progressive disease on fluorouracil based chemotherapy OR
  * Recurrence of disease within 12 months of adjuvant therapy with fluorouracil
* No known CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Granulocyte count greater than 1500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT no greater than 3 times ULN (no greater than 5 times ULN if liver involved)

Renal:

* Creatinine no greater than 2.0 mg/dL
* Calcium no greater than 12.0 mg/dL

Cardiovascular:

* No myocardial infarction within past 6 months
* No congestive heart failure requiring therapy

Neurologic:

* No severe psychiatric disorders
* No history of seizures

Other:

* No active or uncontrolled infection
* HIV negative
* No prior malignancy within past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No uncontrolled diabetes mellitus (random blood sugar 200 mg/dL or greater)
* No other severe concurrent disease
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* Prior oxaliplatin allowed
* No prior irinotecan or topotecan

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent phenytoin, phenobarbital, or other antiepileptic prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 1998-10; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, MD, Study Chair — University of Southern California
Locations (3):
- United States (3):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California